CLINICAL TRIAL: NCT05129683
Title: Effects of a Single Session of Anodal Cerebellar Transcranial Direct Current Stimulation vs Anodal Cerebral Transcranial Direct Current Stimulation on Balance, Mobility and Cognition in Stroke Patients
Brief Title: Single Session of Anodal Cerebellar vs Cerebral Transcranial Direct Current Stimulation in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01141 Qurat Study1
Record Dates: First submitted 2021-09-23; First posted 2021-11-22 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Stroke
Keywords: Transcranial Direct Current Stimulation; Anodal Cerebral
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anodal tDCS cerebellar stimulation group: (Experimental): Anodal tDCS cerebellar stimulation
  Interventions: Other: Anodal tDCS cerebellar stimulation group
- Anodal tDCS cerebral (M1) stimulation group: (Experimental): Anodal tDCS cerebral (M1) stimulation
  Interventions: Other: Anodal tDCS cerebral (M1) stimulation group
- Sham Group (Sham Comparator): Sham: Single-session a-tDCS (2 mA, 20 min),
  Interventions: Other: sham group

INTERVENTIONS:
Other: Anodal tDCS cerebellar stimulation group — Single-session atDCS (2 mA, 20 min). The active (anode) and the returning (cathode) electrodes will be placed bilaterally over the cerebellum (1 -2 cm below inion of occipital bone) and the right buccinator muscle, respectively Xbox kinect based balance and mobility training using games from Xbox Adventure Pack for 50 mins will also be given
  Arms: Anodal tDCS cerebellar stimulation group:
Other: Anodal tDCS cerebral (M1) stimulation group — single session a-tDCS (2 mA, 20 min), the anode will be positioned over the lesioned M1 (C3, International 10-20 system) and the cathode would be located over the supraorbital area. xbox kinect based balance and mobility training using games from Xbox Adventure Pack for 50 mins.
  Arms: Anodal tDCS cerebral (M1) stimulation group:
Other: sham group — single session a-tDCS (2 mA, 20 min), Sham tDCS followed a similar protocol as Anodal tDCS cerebral (M1) stimulation and arrangement but stimulation for 30 s, after which the current was ramped-down and turned off for the rest of the treatment. xbox kinect based balance and mobility training using games from Xbox Adventure Pack for 50 mins.
  Arms: Sham Group

SUMMARY:
To compare the effect of anodal cerebellar transcranial direct current stimulation (ctDCS) vs anodal cerebral direct current stimulation on balance, mobility and cognition in stroke patients in stroke patients

ELIGIBILITY:
Inclusion Criteria:

* ability to give written consent.
* Able to walk unassisted
* Functional status allowing the participants to participate in the balance training.
* Score 6 or above on Johns Hopkins fall risk assessment tool

Exclusion Criteria:

* Neurological diseases, such as Parkinson, Alzheimer
* Any history of psychological illnesses
* Receipt of electrotherapy that might affect the nervous system in the two weeks prior to the study
* Cerebellar disorders
* use of any sedative medicines in the two days prior to the study
* any symptoms of amnesia and depression;
* Memory disorders with scores below 21 on the Mini Mental Status Examination test
* Any signs of severe motor disorders in the lower extremity which cause any movement limitation or deformity
* Any signs of radiculopathy or root lumbar spinal cord involvement
* Any visual or auditory impairment, or vertigo reports
* Use of a heart rate regulator
* Any structural deformities in the lower extremities or the spine
* Any abnormalities in the vestibular system
* History of recent fracture
* Inability to move without assistance

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Changes from the base line, Berg balance scale | Immediately after Intervention and then again after 1 hour.
  Changes from the base line, Immediately after Intervention and then again after 1 hour. The Berg balance scale (BBS) is used to assess the participant's ability to retain stability. The BBS is a widely used test for the assessment of elderly population with impairment of balance and individuals with neurological disorder while sitting, standing, and transferring. This test included both static and dynamic type task. The BBS uses a five-point ordinal scale ranging from 0 (disability) to 4(complete independent performance) and consists of 14 components; the maximum score is 56 points. The scale has been shown to be reliable and valid in stroke patients. A cut-off score of 45 points is used for fall prediction. The BBS involves 14 tasks; a total score of 56. Equipment required for this test were a stop watch or watch with a second's hand and a ruler or other indicator of 2, 5, and 10 inches.
Timed Up and Go test | Immediately after Intervention and then again after 1 hour.
  Changes from the base line, Immediately after Intervention and then again after 1 hour. The Timed Up and Go (TUG) test was designed for the evaluation of balance and Measures mobility in people who are able to walk on their own (assistive device permitted) to find out the risk of fall . The subjects will be required to stand up from a chair, walk 3 m, turn around, return to the chair, and sit down. The time taken to complete this task will be measured. The test will be informed three times. The time required to complete this task will be measured from a stopwatch. The average values from 3 trials, with 1-min rest between each trial, were used for data analysis.
Balance Evaluation Systems Test | Immediately after Intervention and then again after 1 hour.
  Changes from the base line, Immediately after Intervention and then again after 1 hour.. Balance Evaluation Systems Test (BESTest) is a 36-item assessment of balance impairments across 6 postural control contexts. Total score of 108 points total, calculated in to a percentage score (0-100%). Also total sub-scores exist for each above listed system. Item-level scores range from 0 (severe impairment) to 3 (no impairment)

SECONDARY OUTCOMES:
Montreal cognitive Scale | 1 hour
  Changes from the base line, Immediately after Intervention and then again after 1 hour. The tool used for cognitive impairment is Montreal Cognitive Assessment (MoCA). As there is not at all, fairly effective measuring tool for the early diagnosis of cognitive impairments. MoCA is a successful screening test used for the screening of mild cognitive impairment. Scores of MoCA ranges from 0-30.Interpretation of MoCA indicates that score of 26 and above normal, 18 -25 score indicates low cognitive impairments, 10 -18 score considered normal or moderate cognitive impairment while greater than 10 is considered to be severe cognitive impairments.
tDCS Adverse Effects Questionnaire : | Immediately after Intervention and then again after 1 hour.
  Changes from the base line, Immediately after Intervention and then again after 1 hour.. Transcranial Direct-Current Stimulation (tDCS) adverse effects questionaire:
  Do you experience any of the following symptoms or side- effects? Headache, Neck pain, Scalp pain, Tingling, Itching, Burning sensation, Skin redness, Sleepiness, Trouble concentrating, Acute mood change, Others (specify)
  for each symptom patient can give value (1-4) (1, absent; 2,mild; 3, moderate; 4, severe)
  If present: Is this related to tDCS? (1, none ; 2, remote; 3, possible; 4, probable; 5, definite)
6 min walk test: Distance (meters) | Immediately after Intervention and then again after 1 hour.
  Changes from the base line, Immediately after Intervention and then again after 1 hour. 6 min walk test was used to measure Functional capacity. It is a sub maximal exercise test which can aid in assessing functional capacity of patients with cardiopulmonary diseases, in this test we find out the maximum distance in meters which an individual covers in 6 min without any support.
Timed 25-Foot Walk test | Immediately after Intervention and then again after 1 hour.
  Changes from the base line, Immediately after Intervention and then again after 1 hour. Timed 25-Foot Walk (T25-FW) test is a quantitative mobility and leg function performance test based on a timed 25-walk. Two trials will be given to the patient and time will be noted in seconds
Johns Hopkins fall risk assessment Tool | Immediately after Intervention and then again after 1 hour.
  Changes from the base line, Immediately after Intervention and then again after 1 hour. Risk of falling was assessed using the Johns Hopkins Fall Risk Assessment score 13,14 ; a score of less than 6 is considered low risk, 6 to 13 is considered moderate risk, and greater than 13 is considered high risk.
Mini mental state examination (MMSE) | Immediately after Intervention and then again after 1 hour.
  Changes from the base line, Immediately after Intervention and then again after 1 hour. Mini mental state examination (MMSE): used to screen for cognitive impairment in elderly. The maximum MMSE score is 30 points. A score of 20 to 24 suggests mild dementia, 13 to 20 suggests moderate dementia, and less than 12 indicates severe dementia.

CONTACTS AND LOCATIONS:
Overall Officials: Arshad Nawaz Malik, PhD, Principal Investigator — Riphah International University
Locations (1):
- Akbar Hospital, Gujrat, Dhok Gujra, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No